CLINICAL TRIAL: NCT03119090
Title: Cross-sectional Analysis of Non-invasive Measures of Ventricular Systolic and Diastolic Function and Biomarkers in the Fontan Circulation
Brief Title: Fontan Imaging Biomarkers (FIB) Study
Acronym: FIB
Status: Completed | Type: Observational
Sponsor: Boston Children's Hospital (Other)
Collaborators: Evan's Heart Fund (Unknown); Mend a Heart Foundation (Unknown); Matthew Hearts of Hope Foundation (Unknown)
Responsible Party: Principal Investigator, Rahul Rathod, Cardiologist, Boston Children's Hospital
Other Study IDs: IRB-P00017430
Record Dates: First submitted 2017-04-10; First posted 2017-04-18 (Actual); Last update posted 2021-11-05 (Actual); Status verified 2021-11

CONDITIONS: Single-ventricle; Congenital Heart Disease
Keywords: biomarkers; Fontan operation; Single ventricle; congenital heart disease
MeSH Terms: conditions — Univentricular Heart; Heart Defects, Congenital

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood and urine samples are biobanked for current and future study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The goal of the Fontan Imaging Biomarkers (FIB) study is to identify the associations of blood and urine biomarkers to imaging parameters of ventricular mechanics.

DETAILED DESCRIPTION:
This study has the following research questions:

1. What is the reproducibility of ventricular systolic function measurements (including ventricular strain) in Fontan patients using echocardiography (Echo) and cardiac magnetic resonance imaging (CMR)?
2. What is the reproducibility of ventricular diastolic function measurements (including tissue Doppler and strain rate) in Fontan patients using Echo and CMR?
3. Is there a correlation between ventricular function measurements and circulating biomarkers (including galectin-3 levels, NT-proBNP, ST2, and MELD-XI score)?

ELIGIBILITY:
Inclusion Criteria:

* All patients with Fontan circulation undergoing clinically indicated CMR at Boston Children's Hospital will be considered for the study

Exclusion Criteria:

* Inadequate imaging quality to perform proposed analysis
* Patients <15 kg will be excluded to simplify compliance with BCH minimal risk research blood draw volume guidelines (minimal risk is defined as < 5% total blood volume)

Min Age: 3 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients after the Fontan operation
Sampling Method: Non-Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2015-09; Primary Completion 2021-07 (Actual); Study Completion 2021-07 (Actual)

PRIMARY OUTCOMES:
Biomarkers | Through study completion, an average of 3 years
  Correlation of biomarkers and imaging parameters of ventricular mechanics

SECONDARY OUTCOMES:
Diastolic function | Through study completion, an average of 3 years
  Reproducibility of parameters of systolic function
Systolic function | Through study completion, an average of 3 years
  Reproducibility of parameters of systolic function

CONTACTS AND LOCATIONS:
Overall Officials: Rahul H Rathod, MD, Principal Investigator — Boston Children's Hospital
Locations (1):
- Boston Children's Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No